CLINICAL TRIAL: NCT01621763
Title: An Open Label, Balanced, Randomized, Two Treatment, Two Sequence, Two Period, Single-dose, Crossover Oral Bioequivalence Study of Clopidogrel 300 mg Tablets of Dr. Reddy's India and Plavix® 300 mg Tablets Under Fed Conditions
Brief Title: Bioequivalence Study of Clopidogrel Tablets 300 mg Under Fed Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dr. Reddy's Laboratories Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 305-08
Record Dates: First submitted 2012-06-14; First posted 2012-06-18 (Estimated); Last update posted 2012-06-25 (Estimated); Status verified 2008-09

CONDITIONS: Healthy
MeSH Terms: interventions — Clopidogrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Clopidogrel (Experimental): Clopidogrel tablets 300 mg of Dr. Reddy's Laboratories Limited
  Interventions: Drug: Clopidogrel
- Plavix (Active Comparator): Clopidogrel Tablet 300 mg
  Interventions: Drug: Clopidogrel

INTERVENTIONS:
Drug: Clopidogrel — Clopidogrel Tablets 300 mg
  Other Names: Plavix

SUMMARY:
To compare the bioavailability and characterize the pharmacokinetic profile of the Sponsor's formulation (Clopidogrel Bisulfate 300 mg Tablets) with respect to the reference formulation (Plavix® 300 mg tablets) in healthy, adult, human, male subjects under fed conditions and to assess the bioequivalence.

DETAILED DESCRIPTION:
An open label, balanced, randomized, two treatment, two sequence, two period, single-dose, crossover oral bioequivalence study of Clopidogrel Bisulfate 300 mg Tablets of Dr. Reddy's Laboratories Ltd., India and Plavix® (Clopidogrel Bisulfate) 300 mg Tablets of Bristol-Myers Squibb/Sanofi pharmaceuticals partnership Bridgewater, NJ 0880750086441, USA, in healthy, adult, human male subjects under fed conditions.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult human male volunteers between 18 and 55 years of age (both inclusive) living in and around Ahmedabad city of western part of India.
* Having a Body Mass Index (BMI) between 18.5 and 24.9 (both inclusive), calculated as weight in kg/height in m2.
* Not having any significant diseases or clinically significant abnormal findings during screening, medical history, clinical examination, laboratory evaluations, 12-lead ECG and X-ray chest (postero-anterior view) recordings.
* Able to understand and comply with the study procedures, in the opinion of the Principal investigator.
* Able to give voluntary written consent for participation in the trial.

Exclusion Criteria:

* Known hypersensitivity or idiosyncratic reaction to Clopidogrel or any related drug.
* History or presence of any disease or condition which might compromise the haemopoietic, renal, hepatic, endocrine, pulmonary, central nervous, cardiovascular, immunological, dermatological, gastrointestinal or any other body system.
* Ingestion of any medication at any time in 14 days prior to the dosing of Period-I. In any such case subject selection was at the discretion of the Principal Investigator.
* Any history or presence of asthma (including aspirin induced asthma) or nasal polyp or NSAID induced urticaria.
* A recent history of alcoholism (less than 2 years) or daily consumption of moderate (180 mL / day) alcohol use or consumption of alcohol within 48 hours prior to receiving the study medicine.
* The presence of clinically significant abnormal laboratory values including APTT and PT during screening.
* Consumption of grapefruit and/or grapefruit products within 48hrs prior to dosing.
* Use of any recreational drugs or history of drug addiction or testing positive in pre-study drug scans.
* History of psychiatric disorders.
* A history of difficulty in donating blood.
* Donation of blood (1 unit or 350 mL) within 90 days prior to receiving the first dose of IP.

Note: In case the blood loss was less than or equal to 200 mL; subject was enrolled 60 days after blood donation.

* Smokers, who smoked more than 10 cigarettes / day or inability to abstain from smoking during the study.
* A positive hepatitis screen including hepatitis B surface antigen, HCV antibodies.
* A positive test result for HIV antibody and/or syphilis.
* The receipt of an investigational product or participation in a drug research study within a period of 90 days prior to the first dose of study medication. Elimination half-life of the study drug was taken into consideration for inclusion of the subject in the study.

Note: If subject had participated in a study in which blood loss was less than or equal to 200 mL, subject was dosed 60 days after the last sample of previous study.

* An unusual diet, for whatever reason (e.g. low-sodium), for four weeks prior to receiving the study medication and throughout the subjects' participation in the study. In any such case subject selection was at the discretion of the Principal Investigator.
* Any history of peptic ulcer disease, which include gastric & duodenal ulcer or any other bleeding disorders.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2008-09; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Area under curve(AUC) | at pre-dose 0.25, 0.50, 0.75, 1.00, 1.25, 1.50, 1.75, 2.00, 2.25, 2.50, 3.00, 4.00, 6.00, 8.00, 12.00, 16.00, 20.00, 24.00, 36.00 and 48.00 hours post dose

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Dimple Shah, MD, Principal Investigator — Lambda Therapeutic Research Ltd.
Locations (1):
- Lambda Therapeutic Research Ltd, Ahmedabad, Gujarat, India